CLINICAL TRIAL: NCT06182202
Title: Comparing Intact and Residual Amputated Neuromuscular Physiology
Brief Title: Comparing Intact and Residual Amputated Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Carolina State University (Other)
Responsible Party: Principal Investigator, He Huang, Jackson Family Distinguished Professor, North Carolina State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24436
Record Dates: First submitted 2022-07-08; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Amputation
Keywords: Amputees; Electromyography; Ultrasound; Neuromuscular Physiology; Prostheses; Muscle Activation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Individuals Without Amputation (No Intervention): No Intervention Tested in identical tasks for comparison to Individuals with Amputation
- Individuals With Amputation (Experimental): Tasks with a passive prosthesis Tasks with a powered active prosthesis
  Interventions: Device: Powered Prosthesis

INTERVENTIONS:
Device: Powered Prosthesis — Custom in-house powered prosthetic device (used in prior studies, see Citations).
  Arms: Individuals With Amputation

SUMMARY:
Lower limb amputees rely on their prosthetic to remain active and lead an independent life. In recent years, measuring residual muscle activity has been used to interpret a user's intent and thereby modulate prosthesis control. However, little knowledge is held on how residual muscle activity differs from non-amputated muscle. The research team will analyze and compare neuromuscular physiology in non-amputee individuals and amputees' non-amputated and residual muscles across functional tasks to better understand how amputees control their muscles. Such information will inform design of modern prosthesis controllers.

DETAILED DESCRIPTION:
There will be approximately 80 participants in this study: 40 who have lower-limb amputations and 40 who do not.

A minimum of 48 hours will separate each testing session.

A warm-up is incorporated into every session and subjects will regularly take breaks between trials. The research team will check in with them regularly, and they are welcome to tell us when they want a break or stop at any time for any reason.

Subjects will be asked to conducted controlled isolated muscle activity of their ankle muscles, given feedback of their muscle activation to control their effort and prevent fatigue. Following activity of isolated muscles, subjects will be asked to conduct functional tasks including quiet standing, postural sways, sitting down and standing up, squats, heel-raises, and walking.

Individuals with amputation will conduct the tasks with their personal passive prosthesis device as well as a powered active prosthesis (following socket fitting and appropriate adjustment to comfort by a certified, trained prosthetist) to compare muscle activity in functional tasks. Individuals without amputation will conduct the tasks for further comparison.

Surface electromyography, ultrasound, and motion capture data will be used to record muscle activation, muscle architecture, and joint biomechanics respectively and evaluate observations and effects between residual and intact muscles.

More details are below.

-- The following sensors/devices will be attached for the study. The sensors will be fixed via a double-sided adhesive, self-adhesive wraps, or straps. All are easily removable and adjustable for their comfort. Wearing shorts is recommended to simplify the process of adding sensors.

1. Muscle Activation While Sitting (Session 1):

   a. Muscle Activity Sensors: i. Number: 4 ii. Placement: 1 on the front and back of the leg below the knee.
2. Muscle Activation While Sitting (Sessions 2-3):

   a. Muscle Activity Sensors: i. Same as Session 1 b. Joint Dynamics Device: i. Subjects' on-amputated foot will be strapped into a platform that measures how much they are pulling/pushing or moving their ankle. On tasks thinking about activating the phantom limb, the research team will ask participants to match activities with both limbs so that the research team can record what the participants are thinking about with the phantom limb via the non-amputated foot.

   c. Muscle shape sensors: i. Number: 2 ultrasound probes ii. Placement: On the front and back of their leg, switching legs between sessions.
3. Prosthesis Fitting (Sessions 4-6):

   a. Muscle Activity Sensors: i. Same as Session 1 b. Socket: i. A trained prosthetist will cast and fit a socket designed to safely fit the muscle activity sensors.

   c. Powered Prosthesis Device i. A trained prosthetist will assist aligning the casted socket with a powered prosthesis the research team have in the lab.
4. Functional Tasks (Sessions 7-16):

   a. Muscle Activity Sensors: i. Number: 18 ii. Placement: 1 on the front and back of the leg below the knee, 2 on the front of the leg above the knee, 1 on the back of the leg below the knee (5 per leg), 2 on the arm above and below the elbow (4 per arm) b. Socket: i. Fitted in earlier sessions c. Powered Prosthesis Device i. Fitted and aligned in earlier sessions d. Movement measurement markers: i. Number: 40 in total. ii. Placement: 4 on head, 5 on torso, 7 on each arm, 5 on hips, 3 on each leg, 1 on each ankle, toes and heels (on the shoe).

   e. Harness: i. A harness attached to the ceiling will be used to catch subjects case of any fall during the experiment.

During each visit the research team will ask subjects to do all the following:

1. Muscle Activation While Sitting (Sessions 1-3): Come to the lab for 3 initial sessions, where they will:

   1. Practice muscle activation of their ankle muscles while wearing sensors measuring their muscle activity and shape. There will be a brief calibration to their maximum effort to ensure muscle activation will be less than maximum effort throughout the rest of the study.
   2. The research team will provide them with visual biosignal feedback to guide them how to control their muscles.
2. Prosthesis Fitting (Sessions 4-6): Attend a session where a trained prosthetist will cast their residual limb for a socket, followed by 1, 2, or 3 fitting (up to 3 total) sessions with their socket and a powered prosthesis with a certified prosthetist. Each visit will last up to two hours. The prosthetist will duplicate their current socket and ask them to wear it with a powered prosthesis. The prosthetist will also conduct modifications if they do not like the socket to ensure fit and their comfort while wearing the socket.
3. Functional Tasks (Sessions 7-16): Once the fit has been finalized, the participants will come to the lab for up to 10 additional sessions for functional tasks. During each visit, the participants will be asked to practice modulating and controlling the activation of the amputated and non-amputated muscles. After training and practicing activating and controlling the muscles, the research team will then ask the participants to conduct the following tasks:

   1. Quiet standing (not moving)
   2. Postural sway (leaning forward and backward)
   3. Sitting down and standing up repeatedly
   4. Squatting
   5. Standing up on toes (heel-raises)
   6. Walking on a treadmill at their preferred walking speed

Handrails (both left and right) will be always available to allow balance support if needed, and additional harness protection is available.

Individuals without amputation will conduct the functional tasks set once. Individuals with amputation will be asked to do the functional task set both with their passive prosthesis and a powered prosthesis to determine if the powered device improves functional performance, in addition to compare to individuals without amputation. At times, the research team will give them auditory feedback to help the participants time the motion, and visual biosignal feedback to guide them on how the participants place the weight between legs.

The research team expect the participants to come in for up to additional 10 sessions for these activities to account for adaptations in performance when using a powered prosthesis, and post-training evaluations of their amputated and non-amputated muscles. This estimate also accommodates necessary setup and take-down time that subjects must be present for, while maintaining reasonable individual session periods.

ELIGIBILITY:
Inclusion Criteria for Individuals without Amputation:

* Live in the United States
* Are 18 years of age or older
* Can walk across low-level environmental barriers such as curbs, stairs, or uneven surfaces unassisted and without much difficulty

Exclusion Criteria for Individuals without Amputation:

- Have any cognitive, visual, or balance impairments that affects your ability to provide informed consent or to follow instructions during the experiments

* Have had a stroke
* Have heart disease
* Weigh 450 pounds or more (for harness safety)
* Have a girth/waist circumference more than 49 inches (124.4 cm) (for harness safety)
* Have allergies to adhesives

Inclusion Criteria for Individuals with Amputation:

* Live in the United States
* Are a unilateral lower-limb amputee
* Have lower limb length from the knee to where the amputation occurred at least 10cm long
* Can walk across low-level environmental barriers such as curbs, stairs, or uneven surfaces unassisted and without much difficulty

Exclusion Criteria for Individuals with Amputation:

- Have any cognitive, visual, or balance impairments that affects your ability to provide consent or to follow instructions during the experiments

* Have had a stroke
* Have heart disease
* Had skin lesions/incomplete healing following amputation
* Have ulcers
* Have lower limb length from the knee to where the amputation occurred less than 10cm long
* Weigh 450 pounds or more (for harness safety)
* Have a girth/waist circumference more than 49 inches (124.4 cm) (for harness safety)
* Have allergies to adhesives

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Motor Unit Action Potential Amplitudes | Through study completion (an average of 36 months).
  The investigators will measure muscle activity via electromyography on the individuals' muscles controlling their ankle joint (note for residual muscle they are controlling their phantom limb).
  Properties of motor units will be gathered from surface electromyography (EMG) decomposed into individual motor unit firings.
  These properties will be compared between intact and residual muscle.
Motor Unit Coherence | Through study completion (an average of 36 months).
  The investigators will measure muscle activity via electromyography on the individuals' muscles controlling their ankle joint (note for residual muscle they are controlling their phantom limb).
  Properties of motor units will be gathered from surface electromyography (EMG) decomposed into individual motor unit firings.
  These properties will be compared between intact and residual muscle.

SECONDARY OUTCOMES:
Muscle Architecture Properties -- Muscle Volume | Through study completion (an average of 36 months).
  The investigators will measure muscle architecture via ultrasound on the individuals' muscles controlling their ankle joint.
  Properties of architecture will be compared between residual muscle and intact muscle of both participant groups.

CONTACTS AND LOCATIONS:
Locations (1):
- North Carolina State University, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang S, Wensman JP, Ferris DP. Locomotor Adaptation by Transtibial Amputees Walking With an Experimental Powered Prosthesis Under Continuous Myoelectric Control. IEEE Trans Neural Syst Rehabil Eng. 2016 May;24(5):573-81. doi: 10.1109/TNSRE.2015.2441061. Epub 2015 Jun 4. PMID 26057851

DOCUMENTS (1):
  • Informed Consent Form (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT06182202/ICF_000.pdf